CLINICAL TRIAL: NCT00161577
Title: Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety and Efficacy of Ketorolac in the Management of Post-Operative Pain After Heart Surgery
Brief Title: Use of Ketorolac in Management of Post-Operative Pain After Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Gregory Kerr, MD, Weill Cornell Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0903-886
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Pain Management Following Cardiopulmonary Bypass Surgery
Keywords: Ketorolac
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Group A = Ketorolac
  Interventions: Drug: Ketorolac
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketorolac — Intravenous ketorolac every 6 hours for 24 hours
  Other Names: Toradol
  Arms: A
Other: Placebo — Placebo Comparator
  Arms: B

SUMMARY:
This study evaluates the safety and efficacy of ketorolac for post-operative pain management after heart surgery. Ketorolac appears to provide enhanced pain relief while also decreasing the requirements for morphine during the (immediate) 24-hour post-operative period.

DETAILED DESCRIPTION:
Current practice at this institution does not include routine use of ketorolac for post-operative pain management of patients undergoing cardiac surgery. The investigators hypothesize that using Ketorolac as an adjunct to IV morphine can positively impact patient outcomes and reduce the occurrence of possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years of age at the screening visit.
* Undergoing coronary artery bypass graft or single valve repair or replacement requiring cardiopulmonary bypass.
* American Society of Anesthesiology (ASA) Physical Class 3, or 4.
* Willing able to use a PCA Pump
* Willing to receive iv morphine for 24 hours post initial ketorolac dose to control pain.
* Capable of speaking and understanding English sufficiently to provide written informed consent and responses to pain assessment scales and neurological questionnaires.

Exclusion Criteria:

* Allergy or sensitivity to nonsteroidal anti-inflammatory drugs
* History of gastrointestinal bleeding or peptic ulcer
* Serum creatinine = 2.0 mg/dl or rise in serum creatinine of = 0.5 mg/dl or 25% within the preceding 10 days if known with the exception of patients with Dialysis Dependent End Stage Renal Disease (ESRD).
* Hepatic dysfunction
* Patients with low cardiac output syndrome (cardiac index < 2.0) after cardiopulmonary bypass or pre-op ejection fraction < 30%
* Inability to operate PCA pump
* Cardiothoracic reoperations
* Bleeding disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Total morphine administered | 24 hours post operatively

SECONDARY OUTCOMES:
Chest tube drainage | 24 hours post operatively
Respiratory Assessments (NIF, VC) | 24 hours post operatively
VAS Pain Scale | 24 hours post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Gergory Kerr, M.D., MBA, Principal Investigator — Weill Medical College of Cornell University, New York Presbyterian Hospital
Locations (1):
- New York Presbyterian Hospital, Weill Cornell Medical College, New York, New York, United States